CLINICAL TRIAL: NCT00206414
Title: Arimidex/Faslodex/Iressa Study: A Phase II Trial of Primary Systemic Therapy Using a Combination of Arimidex, Faslodex and Iressa (Gefitinib) in Postmenopausal Women With Hormone Receptor Positive Breast Cancer
Brief Title: Arimidex/Faslodex/Iressa Study: A Trial Using Arimidex, Faslodex and Iressa in Women With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty accruing subjects the study accrual was closed
Sponsor: Baylor Breast Care Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-14732
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: BREAST CANCER
Keywords: HORMONE RECEPTOR POSITIVE BREAST CANCER
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Fulvestrant; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iressa Day 1 with Arimidex and Faslodex (Experimental): Subjects randomized to Iressa on Day 1 in combination with Arimidex and Faslodex.
  Interventions: Drug: Iressa Day 1 given with Arimidex and Faslodex
- Iressa Day 21 with Arimidex and Faslodex (Active Comparator): Subjects randomized to Iressa Day 21 in combination with Arimidex and Faslodex
  Interventions: Drug: Iressa Day 21 given with Arimidex and Faslodex

INTERVENTIONS:
Drug: Iressa Day 1 given with Arimidex and Faslodex — timing of administration of iressa is the study factor
  Other Names: gefitinib
  Arms: Iressa Day 1 with Arimidex and Faslodex
Drug: Iressa Day 21 given with Arimidex and Faslodex — Timing of Iressa is the study factor
  Other Names: gefitninb
  Arms: Iressa Day 21 with Arimidex and Faslodex

SUMMARY:
The investigators want to know if combining Arimidex and Faslodex with Iressa will be an effective treatment for breast cancer. They also want to know, using special tests on the tumor, the changes that occur with the treatment so they can try to improve their treatment for breast cancer in the future.

DETAILED DESCRIPTION:
Over the last three decades, a steady shift has occurred in the management of breast cancer. Because it was traditionally viewed as a local disease, many advocated the use of radical surgery to achieve maximum survival benefit. This view has been slowly replaced by a broader biologic view that recognizes the often systemic nature of breast cancer, even when it appears to be localized to the breast. Results from randomized clinical trials have demonstrated that less extensive surgery or lumpectomy plus radiation therapy are optimal for local management of early breast cancer. In addition to the less radical approach to surgical treatment of breast cancer, other randomized clinical trials established the value of postoperative (adjuvant) systemic therapy in improving overall survival by eradicating micrometastatic disease, the major cause of mortality from breast cancer. An improved survival has been shown from using chemotherapy as well as the antiestrogen tamoxifen in the adjuvant setting and has been confirmed through the overview analyses from the Early Breast Cancer Trialist Collaborative Group. Despite the well-documented benefits of adjuvant systemic therapy, it is not effective in preventing death from breast cancer in all patients who are candidates for such treatment. The worth of such therapy can only be judged in retrospect upon disease relapse, a time when breast cancer is nearly always incurable. Currently, there are few reliable methods to predict the success or failure of a particular postoperative treatment modality and better ways to predict and optimize outcome are needed. Preoperative (primary, neoadjuvant) systemic therapy is an alternative approach that is based on a strong rationale. With the tumor still in place and directly accessible, this form of therapy allows direct observation of response to treatment which may predict the likelihood of controlling distant micrometastatic disease and also enables the sampling of tissue to explore molecular correlates of response and also the mechanisms of action of therapeutic agents. Furthermore, it allows early identification of patients with refractory disease who might benefit from alternative treatments before they develop macrometastatic disease and miss the opportunity for a cure. Primary systemic therapy can also help facilitate surgery and debulking of disease in those patients with initially inoperable tumors, as well as improve the odds of breast conservation.

A pivotal trial that established the role of preoperative systemic therapy was the NSABP trial B-187. In this trial, women with localized breast cancer were randomized to receive Adriamycin, Cytoxan (AC) either preoperatively or postoperatively. There was no difference between the two groups in disease-free and overall survival. Furthermore, quantifying tumor response preoperatively allowed prediction of patient outcome in terms of disease-free and overall survival. Specifically, patients achieving a pathologic complete response, i.e., complete disappearance of invasive cancer on pathologic examination, had the best outcome, establishing the role of response as a valid surrogate predictor of the sensitivity of distant micrometastatic disease to chemotherapy and subsequent clinical outcome. In addition, breast-conserving surgery was more frequently performed in the preoperative treatment group, an advantage over the postoperative treatment approach. Most importantly, however, NSABP trial B-18 showed conclusively that primary systemic therapy is safe and does not place patients at a disadvantage by delaying primary surgical treatment. Another large, multicenter prospective trial conducted by the European Organization for Research and Treatment of Cancer (EORTC) confirmed the findings of NSABP trial B-18.

Primary study objective:

* To determine the clinical response rate of primary breast cancer to the combination of Arimidex, Faslodex, and Iressa

Secondary study objectives:

* To study molecular changes in response to treatment
* To determine the pathologic response rate
* To assess the tolerability and safety of the combination regimen

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must be female
2. Postmenopausal status, defined as any one of the following criteria:

   1. documented history of bilateral oophorectomy;
   2. age 60 years or more;
   3. ages 45 to 59 and satisfying one or more of the following criteria:

      * amenorrhea for at least 12 months and intact uterus;
      * amenorrhea for less than 12 months and a follicle stimulating hormone (FSH) concentration within premenopausal range including:

        * patients who have had a hysterectomy;
        * patients who have received hormone replacement.
3. Patients must have histologically confirmed invasive breast cancer with a primary tumor of 3 cm or more in greatest dimension as measured by clinical examination.
4. Estrogen receptor and/or progesterone receptor positive disease
5. Patients must not have received any prior treatment for current or newly diagnosed breast cancer.
6. Patients must have not received previous treatment with any of the study medications or similar drugs.
7. No use of selective estrogen receptor modulators (SERM) such as raloxifene or similar agents in the past 2 years.
8. World Health Organization (WHO) performance status of 0, 1, or 2
9. Adequate organ function defined as follows:

   1. adequate renal function, defined by a serum creatinine within 3 times the upper limits of normal;
   2. adequate liver function, defined by total bilirubin, AST, ALT, and alkaline phosphatase within 3 times the upper limits of normal;
   3. adequate bone marrow function, defined as a white blood cell (WBC) > 3.0 ml, platelet (PLT) > 75,000/ul, hemoglobin (Hb) > 9 gm/l
10. Willing to undergo breast core biopsies as required by the study protocol
11. Ability to understand and sign a written informed consent for participation in the trial
12. Life expectancy of at least 1 year.

Exclusion Criteria:

1. Known severe hypersensitivity to Iressa or any of the excipients of this product
2. Premenopausal status
3. Patients with synchronous bilateral breast cancer
4. Patients with diffuse tumors that cannot be clearly measurable, such as inflammatory breast cancer
5. Other coexisting malignancies with the exception of basal cell carcinoma or cervical cancer in situ
6. Patients with brain metastasis
7. WHO performance status of 3 or 4
8. As judged by the investigator, uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the clinical trial.
10. Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St. John's wort
11. Concurrent treatment with estrogens or progestins. Patients must stop these drugs at least two weeks prior to study entry.
12. Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment
13. Platelet count less than 75,000
14. In the opinion of the investigator, bleeding diathesis or anticoagulation therapy that would preclude intramuscular injections.
15. History of hypersensitivity to castor oil
16. Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded).
17. Patients with recurrent breast cancer. Patients with contralateral second primary breast cancers are eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Primary study objective - To determine the clinical response rate of primary breast cancer to the combination of Arimidex, Faslodex, and Iressa | until disdase progression

SECONDARY OUTCOMES:
Secondary study objectives - To study molecular changes in response to treatment, to determine the pathologic response rate, and to assess the tolerability and safety of the combination regimen | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor Breast Center
Locations (1):
- Baylor Breast Center, Houston, Texas, United States

REFERENCES:
- [Derived] Massarweh S, Tham YL, Huang J, Sexton K, Weiss H, Tsimelzon A, Beyer A, Rimawi M, Cai WY, Hilsenbeck S, Fuqua S, Elledge R. A phase II neoadjuvant trial of anastrozole, fulvestrant, and gefitinib in patients with newly diagnosed estrogen receptor positive breast cancer. Breast Cancer Res Treat. 2011 Oct;129(3):819-27. doi: 10.1007/s10549-011-1679-8. Epub 2011 Jul 27. PMID 21792626
- See also: Web Site — http://www.breastcenter.tmc.edu